CLINICAL TRIAL: NCT06533475
Title: An Open-Label, Randomized Study to Evaluate the Relative Bioavailability of a New Tablet Formulation of Minzasolmin and the Potential Effect of Food on the Pharmacokinetics of Minzasolmin in Healthy Participants
Brief Title: A Study to Assess the Bioavailability of a New Tablet Formulation of Minzasolmin and the Effect of Food in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UP0152; 2024-511301-31-00 (Registry Identifier: EU CT number); U1111-1306-5483 (Other: UTN)
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
Keywords: minzasolmin; Phase 1; Healthy Participants; Bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Treatment A-B-C (Experimental): Participants will be randomized to receive single doses of minzasolmin with and without food on different Days with a 4-day Washout Period between doses. A: Granules in capsule (fasting); B: Tablet formulation (fasting); C: Tablet formulation (fed).
  Interventions: Drug: Minzasolmin tablet formulation under fasting condition; Drug: Minzasolmin Granules in capsule under fasting condition; Drug: Minzasolmin tablet formulation under fed condition
- Treatment B-C-A (Experimental): Participants will be randomized to receive single doses of minzasolmin with and without food on different Days with a 4-day Washout Period between doses. B: Tablet formulation (fasting); C: Tablet formulation (fed); A: Granules in capsule (fasting).
  Interventions: Drug: Minzasolmin tablet formulation under fasting condition; Drug: Minzasolmin Granules in capsule under fasting condition; Drug: Minzasolmin tablet formulation under fed condition
- Treatment C-A-B (Experimental): Participants will be randomized to receive single doses of minzasolmin with and without food on different Days with a 4-day Washout Period between doses. C: Tablet formulation (fed); A: Granules in capsule (fasting); B: Tablet formulation (fasting).
  Interventions: Drug: Minzasolmin tablet formulation under fasting condition; Drug: Minzasolmin Granules in capsule under fasting condition; Drug: Minzasolmin tablet formulation under fed condition
- Treatment A-C-B (Experimental): Participants will be randomized to receive single doses of minzasolmin with and without food on different Days with a 4-day Washout Period between doses. A: Granules in capsule (fasting); C: Tablet formulation (fed); B: Tablet formulation (fasting).
  Interventions: Drug: Minzasolmin tablet formulation under fasting condition; Drug: Minzasolmin Granules in capsule under fasting condition; Drug: Minzasolmin tablet formulation under fed condition
- Treatment B-A-C (Experimental): Participants will be randomized to receive single doses of minzasolmin with and without food on different Days with a 4-day Washout Period between doses. B: Tablet formulation (fasting); A: Granules in capsule (fasting); C: Tablet formulation (fed).
  Interventions: Drug: Minzasolmin tablet formulation under fasting condition; Drug: Minzasolmin Granules in capsule under fasting condition; Drug: Minzasolmin tablet formulation under fed condition
- Treatment C-B-A (Experimental): Participants will be randomized to receive single doses of minzasolmin with and without food on different Days with a 4-day Washout Period between doses. C: Tablet formulation (fed); B: Tablet formulation (fasting); A: Granules in capsule (fasting).
  Interventions: Drug: Minzasolmin tablet formulation under fasting condition; Drug: Minzasolmin Granules in capsule under fasting condition; Drug: Minzasolmin tablet formulation under fed condition

INTERVENTIONS:
Drug: Minzasolmin tablet formulation under fasting condition — Drug: Minzasolmin Pharmaceutical form: Tablet formulation under fasting condition
  Other Names: UCB0599
Drug: Minzasolmin Granules in capsule under fasting condition — Drug: Minzasolmin Pharmaceutical form: Granules in capsule under fasting condition
  Other Names: UCB0599
Drug: Minzasolmin tablet formulation under fed condition — Drug: Minzasolmin Pharmaceutical form: Tablet formulation under fed condition
  Other Names: UCB0599

SUMMARY:
The purpose of the study is to estimate the relative bioavailability of a new minzasolmin tablet formulation versus reference 'granules in capsule' formulation in healthy participants and to evaluate the effect of food with the new tablet formulation on the pharmacokinetics (PK) of minzasolmin.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive at the time of signing the informed consent form (ICF)
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Body weight within 45 to 100kg (female) and 50 to 100kg (male) and body mass index (BMI) within the range 18 to 30kg/m2 (inclusive).

Exclusion Criteria:

* Participant has a history of chronic alcohol abuse (more than 24g [males] or 12g [females] per day; 12g pure alcohol are contained in approximately 300mL of beer (5%), 1 small glass [125 mL] of wine [12%], or 1 measure [40mL] of spirits [37.5%]) or drug abuse within the last 1 year from Screening, as defined according to the Diagnostic and Statistical Manual of Mental Disorders
* Study participant has received or intends to use any prescription or nonprescription medicines, including enzyme inhibitors or inducers, any gastric pH modifying agents, over the counter remedies, herbal and dietary supplements (including St. John's Wort) up to 2 weeks (4 weeks for enzyme inducers) or 5 half-lives of the respective drug (whichever is longer) before the first administration of minzasolmin
* Participant has participated in another study of an investigational medicinal product (IMP) (and/or an investigational device) within the previous 30 days or 5 half-lives, whichever is greatest, or is currently participating in another study of an IMP (and/or an investigational device)
* Participant has alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) >1.0x upper limit of normal (ULN)
* Participant has total bilirubin >1.0xULN. Bilirubin >ULN and ≤1.5xULN is acceptable if fractioned and direct bilirubin <35%, and if a baseline diagnosis of Gilbert's syndrome is understood and recorded in ClinBase
* Participant has any clinically relevant electrocardiogram (ECG) finding at the Screening Visit or at Baseline, or a family history of sudden death due to long QT syndrome which, in the opinion of the investigator, would put the participant at increased risk of QT prolongation during the study

In addition, any study participant with any of the following findings will be excluded at Screening:

* QT interval corrected for heart rate using Fridericia's formula >450 msec for males and >470msec for females
* other conduction abnormalities (defined as pulse rate [PR] interval ≥220ms)
* irregular rhythm other than sinus arrhythmia or occasional, rare supraventricular, and rare ventricular ectopic beats

  - Study participant has a medical history or current diagnosis of renal impairment and/or Screening laboratory results show:
* An estimated glomerular filtration rate <90 mL/min/1.73m2 (using the Chronic Kidney Disease Epidemiology Collaboration formula)
* An albumin/creatinine ratio ≥30mg/mmol
* Urinary tract infection; in this case a study participant can be rescreened once the infection has been resolved - Participant has donated blood or experienced blood loss >350mL within the last 1 month before the first IMP administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-09-06 (Actual); Primary Completion 2024-11-17 (Actual); Study Completion 2024-11-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Up0152 1001, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in September 2024 and concluded in November 2024.
Pre-assignment Details: The Participant Flow refers to the Randomized Set.
Groups:
- Treatment ABC: Participants received minzasolmin granules in capsules, administered under fasting conditions (Treatment A) in Period 1 followed by a single dose of minzasolmin tablet under fasting conditions (Treatment B) in Period 2, further followed by a single dose of minzasolmin tablet under fed conditions (Treatment C) in Period 3. Each treatment period was of 1 Day (Days 1, 6, and 11 respectively) only, separated by 4-Days Washout period.
- Treatment BCA: Participants received a single dose of minzasolmin tablet under fasting conditions (Treatment B) in Period 1 followed by a single dose of minzasolmin tablet under fed conditions (Treatment C) in Period 2, further followed by minzasolmin granules in capsules, administered under fasting conditions (Treatment A) in Period 3. Each treatment period was of 1 Day (Days 1, 6, and 11 respectively) only, separated by 4-Days Washout period.
- Treatment CAB: Participants received a single dose of minzasolmin tablet under fed conditions (Treatment C) in Period 1 followed by minzasolmin granules in capsules administered under fasting conditions (Treatment A) in Period 2, further followed by a single dose of minzasolmin tablet under fasting conditions (Treatment B) in Period 3. Each treatment period was of 1 Day (Days 1, 6, and 11 respectively) only, separated by 4-Days Washout period.
- Treatment ACB: Participants received minzasolmin granules in capsules, administered under fasting conditions (Treatment A) in Period 1 followed by a single dose of minzasolmin tablet under fed conditions (Treatment C) in Period 2, further followed by a single dose of minzasolmin tablet under fasting conditions (Treatment B) in Period 3. Each treatment period was of 1 Day (Days 1, 6, and 11 respectively) only, separated by 4-Days Washout period.
- Treatment BAC: Participants received a single dose of minzasolmin tablet under fasting conditions (Treatment B) in Period 1 followed by minzasolmin granules in capsules, administered under fasting conditions (Treatment A) in Period 2, further followed by a single dose of minzasolmin tablet under fed conditions (Treatment C) in Period 3. Each treatment period was of 1 Day (Days 1, 6, and 11 respectively) only, separated by 4-Days Washout period.
- Treatment CBA: Participants received a single dose of minzasolmin tablet (Treatment C) under fed conditions in Period 1 followed by a single dose of minzasolmin tablet (Treatment B) under fasting conditions in Period 2, further followed by minzasolmin granules in capsules (Treatment A), administered under fasting conditions in Period 3. Each treatment period was of 1 Day (Days 1, 6, and 11 respectively) only, separated by 4-Days Washout period.
Period: Overall Study
Arm/Group | Treatment ABC | Treatment BCA | Treatment CAB | Treatment ACB | Treatment BAC | Treatment CBA
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the SS which consisted of all study participants who were randomized and received full or partial study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment ABC | Treatment BCA | Treatment CAB | Treatment ACB | Treatment BAC | Treatment CBA | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (3.6) | 38.0 (6.0) | 44.3 (7.1) | 48.0 (7.5) | 40.7 (8.1) | 43.7 (8.1) | 42.8 (6.6)
Age, Customized [Count of Participants; unit: Participants]
  18 - <65 years | 3 | 3 | 3 | 3 | 3 | 3 | 18
  65 - <85 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=85 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 0 | 2 | 3 | 7
  Male | 2 | 3 | 2 | 3 | 1 | 0 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 3 | 3 | 3 | 3 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 2 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to t (AUC[0-t]) for Minzasolmin
Description: AUC0-t was defined as the area under the plasma concentration-time curve from time zero to the last measurable drug concentration sampling time for Minzasolmin.
Time Frame: Predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, and 96 hour (h) post dose on Day 1, Day 6, and Day 11
Population: The Pharmacokinetics (PK) Set consisted of all study participants in the safety set (SS) who had at least 1 observable PK concentration data point and who had no important protocol deviations affecting the PK during the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms per milliliter (h*ng/mL)
Groups:
- Minzasolmin Capsule (Fasted): All participants who received minzasolmin granules in capsules (Treatment A), administered under fasting conditions in Period 1, 2 and 3. Each treatment period was of 1 Day (Day 1, 6 and 11 respectively) only, separated by 4-Days Washout period.
- Minzasolmin Tablet (Fasted): All participants who received a single dose of minzasolmin tablet (Treatment B) under fasting conditions in Period 1, 2 and 3. Each treatment period was of 1 Day (Day 1, 6 and 11 respectively) only, separated by 4-Days Washout period.
- Minzasolmin Tablet (Fed): All participants who received a single dose of minzasolmin tablet (Treatment C) under fed conditions in Period 1, 2 and 3. Each treatment period was of 1 Day (Day 1, 6 and 11 respectively) only, separated by 4-Days Washout period.
Arm/Group | Minzasolmin Capsule (Fasted) | Minzasolmin Tablet (Fasted) | Minzasolmin Tablet (Fed)
Number analyzed (Participants) | 18 | 18 | 18
hour*nanograms per milliliter (h*ng/mL) | 5612 (34.6) | 5710 (35.5) | 6140 (34.2)
Statistical Analysis 1: Comparison: Minzasolmin Capsule (Fasted) vs Minzasolmin Tablet (Fasted); Test type: Other; GLSM Ratio = 1.018, 90% CI 2-sided [0.9624 to 1.076] — The GLSM ratio was calculated: Minzasolmin tablet (Fasted)/ Minzasolmin Capsule (Fasted)
Statistical Analysis 2: Comparison: Minzasolmin Tablet (Fasted) vs Minzasolmin Tablet (Fed); Test type: Other; GLSM Ratio = 1.075, 90% CI 2-sided [1.024 to 1.130] — The GLSM ratio was calculated as: Minzasolmin Tablet (Fed)/Minzasolmin Tablet (Fasted)

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Zero to Infinity for Minzasolmin
Description: AUC was defined as the area under the plasma concentration-time curve from time zero to infinity for Minzasolmin.
Time Frame: Predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, and 96 h post dose on Day 1, Day 6, and Day 11
Population: The PK set consisted of all study participants in the SS who had at least 1 observable PK concentration data point and who had no important protocol deviations affecting the PK during the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Minzasolmin Capsule (Fasted) | Minzasolmin Tablet (Fasted) | Minzasolmin Tablet (Fed)
Number analyzed (Participants) | 18 | 18 | 18
h*ng/mL | 5656 (34.3) | 5769 (35.5) | 6190 (33.9)
Statistical Analysis 1: Comparison: Minzasolmin Capsule (Fasted) vs Minzasolmin Tablet (Fasted); Test type: Other; GLSM Ratio = 1.020, 90% CI 2-sided [0.9649 to 1.078] — The GLSM ratio was calculated as: Minzasolmin tablet (Fasted)/ Minzasolmin Capsule (Fasted)
Statistical Analysis 2: Comparison: Minzasolmin Tablet (Fasted) vs Minzasolmin Tablet (Fed); Test type: Other; GLSM Ratio = 1.073, 90% CI 2-sided [1.021 to 1.127] — The GLSM ratio was calculated as: Minzasolmin Tablet (Fed)/Minzasolmin Tablet (Fasted)

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Minzasolmin
Description: Cmax was defined as the maximum (peak) observed drug concentration following a single dose administration of Minzasolmin.
Time Frame: Predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, and 96 h post dose on Day 1, Day 6, and Day 11
Population: PK set consisted of all study participants in the SS who had at least 1 observable PK concentration data point and who had no important protocol deviations affecting the PK during the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per mililiter (ng/mL)
Arm/Group | Minzasolmin Capsule (Fasted) | Minzasolmin Tablet (Fasted) | Minzasolmin Tablet (Fed)
Number analyzed (Participants) | 18 | 18 | 18
nanograms per mililiter (ng/mL) | 627.2 (45.9) | 612.9 (54.8) | 622.5 (30.9)
Statistical Analysis 1: Comparison: Minzasolmin Capsule (Fasted) vs Minzasolmin Tablet (Fasted); Test type: Other; GLSM Ratio = 0.9771, 90% CI [0.7966 to 1.199] — The GLSM ratio was calculated as: Minzasolmin tablet (Fasted)/ Minzasolmin Capsule (Fasted)
Statistical Analysis 2: Comparison: Minzasolmin Tablet (Fasted) vs Minzasolmin Tablet (Fed); Test type: Other; GLSM Ratio = 1.016, 90% CI 2-sided [0.7940 to 1.299] — The GLSM ratio was calculated as: Minzasolmin tablet (Fed)/ Minzasolmin tablet (Fasted)

4. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were all AEs starting on or after the date/time of first treatment and up to including 4 days after last treatment, or any unresolved event already present before administration of treatment that worsens in intensity following exposure to the treatment.
Time Frame: From Baseline to end of Safety Follow-Up, up to 48 days
Population: The SS consisted of all study participants who were randomized and received full or partial study medication. Study participants were classified according to the treatment that participants actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Minzasolmin Capsule (Fasted) | Minzasolmin Tablet (Fasted) | Minzasolmin Tablet (Fed)
Number analyzed (Participants) | 18 | 18 | 18
percentage of participants | 16.7 | 22.2 | 22.2

5. Secondary Outcome: Percentage of Participants With Serious Treatment-emergent Adverse Events (TEAEs)
Description: An SAE was defined as any untoward medical occurrence that, at any dose, met 1 or more of the criteria listed:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Important medical events such as (but not limited to) invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias, convulsions not resulting in hospitalization, or development of intervention dependency or intervention abuse.
Time Frame: From Baseline to end of Safety Follow-Up, up to 48 days
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Groups:
- Minzasolmin Tablet (Fed): All participants who received a single dose of minzasolmin tablet (Treatment C) under fed conditions on Day 1 in Period 1, Day 6 in Period 2 and Day 11 in Period 11. Each treatment period was of 1 Day (Days 1, 6, and 11 respectively) only, separated by 4-Days Washout period.
Arm/Group | Minzasolmin Capsule (Fasted) | Minzasolmin Tablet (Fasted) | Minzasolmin Tablet (Fed)
Number analyzed (Participants) | 18 | 18 | 18
percentage of participants | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With TEAEs Leading to Withdrawal From Study
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were all AEs starting on or after the date/time of first treatment and up to including 4 days after last treatment, or any unresolved event already present before administration of treatment that worsens in intensity following exposure to the treatment. Percentage of participants with TEAEs leading to withdrawal from study were reported.
Time Frame: From Baseline to end of Safety Follow-Up, up to 48 days
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Groups:
- MinzasolminTablet (Fed): All participants who received a single dose of minzasolmin tablet (Treatment C) under fed conditions in Period 1, 2 and 3. Each treatment period was of 1 Day (Day 1, 6 and 11 respectively) only, separated by 4-Days Washout period.
Arm/Group | Minzasolmin Capsule (Fasted) | Minzasolmin Tablet (Fasted) | MinzasolminTablet (Fed)
Number analyzed (Participants) | 18 | 18 | 18
percentage of participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline to end of Safety Follow-Up, up to 48 days
Description: A TEAE was defined all AEs starting on or after the date/time of first treatment and up to including 4 days after last treatment, or any unresolved event already present before administration of treatment that worsens in intensity following exposure to the treatment.
Arm/Group | Minzasolmin Capsule (Fasted) | Minzasolmin Tablet (Fasted) | Minzasolmin Tablet (Fed)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 3/18 | 4/18 | 4/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minzasolmin Capsule (Fasted) (N=18) | Minzasolmin Tablet (Fasted) (N=18) | Minzasolmin Tablet (Fed) (N=18)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT06533475/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/75/NCT06533475/SAP_001.pdf